CLINICAL TRIAL: NCT02538562
Title: HER2 Advanced Gastric Epidemiology Study in Korea: An Assessment of HER2 Status in Tumor Tissue Samples of Gastric and Gastro-esophageal (GE) Junction Cancer
Brief Title: Human Epidermal Growth Factor Receptor 2 (HER2) Advanced Gastric Epidemiology Study in Korea
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25697
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 2000 tumor tissue samples will be obtained from 17 local laboratories in Korea. Because the study itself is noninterventional, samples must have been previously collected in accordance with routine clinical practice.

GROUPS / COHORTS (1):
- Study Population: Available tumor samples from patients with gastric or gastroesophageal junction cancer will be analyzed. No study visits or interventions are planned.

SUMMARY:
This study is designed to gather epidemiological data in Korea on HER2 incidence in gastric and gastroesophageal junction cancer as assessed by local laboratories in a real-life setting. No investigational products will be provided or evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Formalin-fixed, paraffin-embedded tumor tissue samples with histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction with locally advanced, recurrent, and/or metastatic disease
* Sufficient invasive tumor tissue for HER2 evaluation, including surgical excision specimens or at least 6 to 8 available biopsies

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Available tumor samples from patients with gastric or gastroesophageal junction cancer will be analyzed. No study visits or interventions are planned.
Sampling Method: Non-Probability Sample
Enrollment: 1695 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2013-04-19 (Actual); Study Completion 2013-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of HER2 positivity among gastric and gastroesophageal junction tumor samples | Up to 12 months of sample collection

SECONDARY OUTCOMES:
Correlation between HER2 status and tumor stage | Up to 12 months of sample collection
Correlation between HER2 status and tumor type | Up to 12 months of sample collection
Correlation between HER2 status and cancer diagnosis | Up to 12 months of sample collection
Correlation between HER2 status and age | Up to 12 months of sample collection
Correlation between HER2 status and gender | Up to 12 months of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- South Korea (14):
  - Dongnam Inst.of Radiological & Medical Sciences, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje university Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan University Hospital, Busan
  - Samsung Changwon Hospital, Changwon
  - Dankook University Hospital, Chungcheongnam-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Yeungnam Univ. Hospital, Daegu
  - Chosun University Hospital, Gwangju
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gyeongsang National University Hospital, Gyeongsangnam-do
  - Chonbuk National Uni Hospital, Jeollabuk-do